CLINICAL TRIAL: NCT00699257
Title: A Prospective, Non-controlled, Clinical Investigation of the Oxford® Partial Knee System
Brief Title: A Clinical Investigation of the Oxford® Partial Knee System
Status: Terminated | Type: Observational
Sponsor: Biomet Orthopedics, LLC (Industry)
Responsible Party: Sponsor
Organization: Zimmer Biomet (Industry)
Other Study IDs: Biomet 12380-63
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis
Keywords: Partial Knee Arthroplasty; Partial Knee Replacement; Arthritis of Medial Compartment of the Knee; Oxford Knee
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Oxford® Partial Knee System

SUMMARY:
The purpose of this prospective data collection is to document the performance and clinical outcomes of the Oxford® Partial Knee System.

ELIGIBILITY:
Inclusion Criteria:

* For use in individuals with osteoarthritis or avascular necrosis limited to the medial compartment of the knee. The implant is intended to be implanted with bone cement.

Exclusion Criteria:

* Infection
* Use in the lateral compartment of the knee
* Rheumatoid arthritis or other forms of inflammatory joint disease
* Revision of a failed prosthesis, failed upper tibial osteotomy or post-traumatic arthritis after tibial plateau fracture
* Insufficiency of the collateral, anterior, or posterior cruciate ligaments which would preclude stability of the device
* Disease or damage to the lateral compartment of the knee
* Uncooperative patient or patient with neurologic disorders who is incapable of following directions
* Osteoporosis
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Distant foci of infections which may spread to the implant site
* Rapid joint destruction, marked bone loss, or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy, neuromuscular disease
* Incomplete or deficient soft tissue surrounding the knee
* Charcot's disease
* A fixed varus deformity (not passively correctable) of greater than 15 degrees
* A flexion deformity greater than 15 degrees

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that have already made the decision to undergo knee surgery and will receive the Oxford® Partial Knee System.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2004-07; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Knee Society Score | 6 weeks, 3 months, 1 year, 3 years, 5 years
Oxford-12 Self Assessment Form | 6 weeks, 3 months, 1 year, 3 years, 5 years

SECONDARY OUTCOMES:
Incidence of revisions and removals | Any time

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Beres, MD, Study Director — Clinical Research, Biomet Orthopedics, LLC